CLINICAL TRIAL: NCT07290920
Title: Sensorimotor Integration in Patients With Tourette Syndrome: an Observational Study.
Brief Title: Sensorimotor Integration in Patients With Tourette Syndrome
Acronym: ISM
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: ISM_L3053
Record Dates: First submitted 2025-12-04; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Tourette Disorder; Sensory Gating
Keywords: Tourette Syndrome; Sense of agency; Sensorimotor integration; Sensory attenuation; Motor control; Predictive processing
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tourette Syndrome Patients: Patients affected by Tourette Syndrome
- Healthy controls: Individuals without neurological or psychiatric disorders

SUMMARY:
The present study investigates the mechanisms underlying the sense of agency in patients with Tourette Syndrome (TS). Previous research has shown that individuals with TS display impairments in both explicit and implicit aspects of agency, possibly due to altered integration between sensory feedback and motor predictions. To explore this hypothesis, the study will examine the phenomenon of sensory attenuation, a marker of sensorimotor integration that has not yet been investigated in this population. Furthermore, the study will assess how alterations in sensorimotor integration are related to the severity of TS symptoms.

DETAILED DESCRIPTION:
The present study aims to investigate the mechanisms underlying the sense of agency in patients with Tourette Syndrome (TS). Previous evidence indicates that individuals with TS exhibit abnormalities in both explicit and implicit (absent intentional binding) experiences of agency. According to a recent theoretical framework, such alterations may stem from impaired sensorimotor integration - specifically, a dysfunction in the ability to combine sensory feedback with motor predictions about the consequences of one's own actions. This deficit may not only affect motor control but also the awareness of self-generated movements, thereby compromising the distinction between self-produced and externally produced actions.

To test this hypothesis, the study will employ the Force Matching Task (FMT), a well-established paradigm used to assess sensory attenuation - the reduced perception of intensity for self-generated sensations compared to externally generated ones. In this task, participants are asked to reproduce a force applied to their finger either by pressing directly with their own finger (self-generated condition) or by controlling a mechanical device (externally generated condition). In healthy individuals, self-generated forces are typically perceived as weaker due to predictive motor mechanisms. A reduced or absent sensory attenuation effect would indicate altered sensorimotor integration.

The primary aim of the study is therefore to evaluate whether patients with Tourette Syndrome show atypical sensory attenuation compared to healthy controls, as an index of altered sensorimotor integration underlying the sense of agency. The secondary aim is to examine the relationship between the degree of sensory attenuation and clinical symptom severity, to determine whether deficits in sensorimotor integration are associated with the intensity of tic expression or other clinical features of the disorder.

ELIGIBILITY:
Inclusion Criteria:

For Tourette Syndrome group:

* Clinical diagnosis of Tourette Syndrome (TS) according to DSM-5 criteria
* Age between 18 and 65 years
* Ability to understand and comply with study procedures
* Written informed consent provided

For Healthy Control group:

* No current or past history of neurological or psychiatric disorders
* Age between 18 and 65 years
* Matched to the TS group for age, sex, and education level
* Ability to understand and comply with study procedures
* Written informed consent provided

Exclusion Criteria:

* History of significant neurological disorders (e.g., brain injury or dementia) or major psychiatric disorders (with the exception of conditions commonly associated with Tourette Syndrome, such as Obsessive-Compulsive Disorder, ADHD, depression, and anxiety);
* Failure or refusal to provide written informed consent;
* Confirmed pregnancy (self-reported) and/or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include adult participants aged 18 to 65 years, comprising two groups: individuals diagnosed with Tourette Syndrome (TS) and healthy control participants. The Tourette group will consist of patients meeting DSM-5 diagnostic criteria for Tourette Syndrome, recruited through specialized neurological and neuropsychiatric clinics. Healthy controls will be recruited from the general population and will be matched to the TS group for age, sex, and education level.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Magnitude of sensory attenuation (difference between self-generated and externally generated force reproduction) | Day 1
  Sensory attenuation

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delorme C, Salvador A, Voon V, Roze E, Vidailhet M, Hartmann A, Worbe Y. Illusion of agency in patients with Gilles de la Tourette Syndrome. Cortex. 2016 Apr;77:132-140. doi: 10.1016/j.cortex.2016.02.003. Epub 2016 Feb 17. PMID 26963083
- [Background] Zapparoli L, Seghezzi S, Zirone E, Guidali G, Tettamanti M, Banfi G, Bolognini N, Paulesu E. How the effects of actions become our own. Sci Adv. 2020 Jul 1;6(27):eaay8301. doi: 10.1126/sciadv.aay8301. Print 2020 Jul. PMID 32937445
- [Background] Brown H, Adams RA, Parees I, Edwards M, Friston K. Active inference, sensory attenuation and illusions. Cogn Process. 2013 Nov;14(4):411-27. doi: 10.1007/s10339-013-0571-3. Epub 2013 Jun 7. PMID 23744445